CLINICAL TRIAL: NCT02569593
Title: Evaluation of the Absorption Rate From Different Oral Fe-supplements in Obese Volunteers Pre- and Post-RYGB: an Interventional Study
Brief Title: Evaluation of the Absorption Rate From Different Oral Fe-supplements in Obese Volunteers Pre- and Post-RYGB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Ina Gesquiere, PharmD-PhD, KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IAS15; s58442 (Other: Clinical Trial Center UZ)
Record Dates: First submitted 2015-10-05; First posted 2015-10-07 (Estimated); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Iron-Dextran Complex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RYGB-patient (Other): Patients with a planned RYGB at UZ Leuven will be recruited. Iron supplements, more specific Ferrodyn and Vista Ferrum will be administrated in these patients before and 1, 3, 6 and 12 months post-RYGB with at least 7 days between the administration of the different supplements.
  Interventions: Dietary Supplement: Iron supplements, more specific Ferrodyn and Vista Ferrum

INTERVENTIONS:
Dietary Supplement: Iron supplements, more specific Ferrodyn and Vista Ferrum — Ferrodyn is an Fe-chelate supplement. One tablet contains 28 mg elemental iron. Vista Ferrum is an iron(II)sulfate supplement. One tablet also contains 28 mg elemental iron. The volunteers will be asked to take the provided supplement orally with 150 mL of water.

SUMMARY:
Obese volunteers who have scheduled a gastric bypass (RYGB) in UZ Leuven will be asked to participate in a cross-over study using commercial available iron supplements. The aim of this study is to evaluate the absorption rate of different oral iron supplements in volunteers before and after RYGB (1, 3, 6 and 12 months post-RYGB).

DETAILED DESCRIPTION:
Patients who met the criteria will be invited to come to the clinical research center at 10 occasions (two times before and 1, 3, 6 and 12 months after RYGB). During each visit the following information will be collected:

* General information concerning sociodemographic and medical background
* The medical history
* Anthropometric measures
* Physical activity by questionnaire
* Food frequency by questionnaire
* Information about menstrual blood loss.

Following an overnight fast, subjects will come to the clinical research center. An intravenous catheter will be inserted to collect blood samples. Before the oral administration, blood samples will be collected for the determination of the serum concentration of different iron status markers. The volunteers will receive first an iron(II)sulfate supplement, followed by a Fe-chelate supplement (at least 7 days between both supplements). After the administration of the supplement, blood samples will be taken at various time points to determine the amount of iron absorption and to investigate if there are any changes in the iron metabolism (at 15, 30, 60, 90 minutes and 2; 2.5; 3; 3.5; 4 and 5 hours after oral administration). There will be a one-week washout period between the tests with each iron supplement. The volunteers will be asked to repeat the test before surgery and 1, 3, 6 and 12 months after surgery for each iron supplement.

ELIGIBILITY:
Inclusion Criteria:

* Obese patients who have planned a RYGB surgery in the University Hospital Leuven
* Low iron status at the preoperative consultation (ferritin < 30 µg/L and/or transferrin saturation <20%)

Exclusion Criteria:

* Patients with a bariatric surgery history
* Smokers (> 15 cigarettes/day)
* Pregnant women
* Lactating women
* Patients with a positive helicobacter pylori screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-12 (Estimated); Study Completion 2018-08

PRIMARY OUTCOMES:
The absorption rate from different oral Fe-supplements | One year
  The rate and extent of absorption of iron wille be estimated by changes in serum iron concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Bart Van der Schueren, Principal Investigator — KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Belgium